CLINICAL TRIAL: NCT02751736
Title: The Effect Of Probiotics From Kimchi (CJLP243) On Bowel Function Restoration After Ileostomy Closure In Patients With Rectal Cancer: A Pilot Randomized Controlled Trial
Brief Title: The Effect Of Probiotics On Bowel Function Restoration After Ileostomy Closure In Patients With Rectal Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Seoul National University Hospital (Other)
Collaborators: HK inno.N Corporation (Industry)
Responsible Party: Principal Investigator, Heung-Kwon Oh, Clinical Associate Professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B-1603-339-003
Record Dates: First submitted 2016-04-07; First posted 2016-04-26 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2017-04

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): * 2 g sachet (CJLP 243) once a day for 3 weeks
  * 10 billion lactic acid bacteria(lactobacillus plantarum CJLP243), maltodextrin, glucose(anhydrous)
  Interventions: Dietary Supplement: CJLP243
- Control (Placebo Comparator): * 2g sachet (near identically appearing placebo) once day for 3 weeks
  * maltodextrin, glucose(anhydrous)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: CJLP243 — Perioperative administration till postoperative weeks 3
  Arms: Intervention
Dietary Supplement: Placebo — Perioperative administration till postoperative weeks 3
  Arms: Control

SUMMARY:
The study will investigate whether Probiotics(CJLP243) given just before and after ileostomy repair operation in patient with rectal cancer improve a bowel function.

ELIGIBILITY:
Inclusion Criteria:

* Age: 20-75
* with rectal cancer
* s/p low anterior resection (double stapled anastomosis)

Exclusion Criteria:

* Metastatic cancer
* Pregnancy
* Valvular heart disease
* s/p intersphincteric resection (index surgery)
* h/o anastomotic leakage (index surgery)
* medically unfit (cardiopulmonary dysfunction, sepsis etc)

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-04; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Memorial Sloan Kettering Cancer Center bowel function index | Postoperative weeks 3
  Subscale: frequency score
Low Anterior Resection Syndrome score | Postoperative weeks 3

SECONDARY OUTCOMES:
Memorial Sloan Kettering Cancer Center bowel function index | Postoperative week 1
Low Anterior Resection Syndrome score | Postoperative week 1
Change of bowel functions index | Between postoperative week 1 to 3
EORTC C30 | Postoperative week 1 and 3
EORTC CR (Colorectal) 29 | Postoperative week 1 and 3
Postoperative complication | till Postoperative weeks 3

IPD SHARING:
Plan to Share IPD: No